CLINICAL TRIAL: NCT04856189
Title: A Phase Ib/II Study of Selinexor Plus Pembrolizumab in Cisplatin-Ineligible or Cisplatin-Refractory Patients With Advanced Urothelial Carcinoma
Brief Title: Selinexor and Pembrolizumab for the Treatment of Cisplatin-Ineligible or Cisplatin-Refractory Locally Advanced or Metastatic Urothelial Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual.
Sponsor: Mamta Parikh (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mamta Parikh, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#289; NCI-2021-02845 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#289 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Refractory Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (selinexor, pembrolizumab) (Experimental): Patients receive selinexor PO on days 1, 8 and 15, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Selinexor

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio

SUMMARY:
This phase Ib/II trial finds the best dose of selinexor and its effect with pembrolizumab in treating patients with urothelial carcinoma that are not eligible to receive the chemotherapy drug cisplatin, or have been given cisplatin and the cancer has gotten worse. Patients must also have urothelial carcinoma that has spread locally, near where it started (locally advanced), or has spread to other parts of the body (metastatic). Selinexor may stop the growth of tumor cells by blocking a protein, called XPO1, that is needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving selinexor and pembrolizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of selinexor in combination with standard-dose pembrolizumab in patients with advanced urothelial carcinoma who are cisplatin-ineligible or platinum-refractory. (Phase Ib) II. To determine the objective response rate (ORR) of selinexor in combination with pembrolizumab in patients with advanced urothelial carcinoma who are cisplatin-ineligible or platinum-refractory. (Phase II)

SECONDARY OBJECTIVES:

I. To further evaluate the toxicity profile of the combination of selinexor with pembrolizumab in patients with advanced urothelial carcinoma.

II. To further evaluate the efficacy of the combination of selinexor with pembrolizumab in patients with advanced urothelial carcinoma as defined by progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed locally advanced or metastatic urothelial carcinoma by histology
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Not eligible to receive cisplatin-based chemotherapy due to renal dysfunction (defined as creatinine clearance [CrCl] =< 60 mL/min), > grade 2 peripheral neuropathy, or ototoxicity (defined as >= grade 2 hearing loss); OR unwillingness of patient to receive cisplatin; OR progressed on one platinum-based chemotherapy regimen for advanced disease
* May have had neoadjuvant or adjuvant platinum-based chemotherapy or intravesical therapy in the past
* >= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1 × 10^9/L
* Platelet count >= 75 × 10^9/L (patients for whom <50% of bone marrow nucleated cells are plasma cells) or >= 50,000/mm3 (patients for whom >= 50% of bone marrow nucleated cells are plasma cells)
* Hemoglobin >= 9 g/dL (may have been transfused)
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) range (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 x ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =< 2.5 x ULN, or AST and ALT levels =< 5 x ULN (for subjects with documented metastatic disease to the liver)
* Creatinine clearance >= 30 mL/min by Cockcroft-Gault formula
* Subjects with active hepatitis B virus (Hep B) are allowed if antiviral therapy for hepatitis B has been given for > 8 weeks and viral load is < 100 IU/mL prior to first dose of trial treatment. Subjects with untreated hepatitis C virus (HCV) are allowed. Subjects with human immunodeficiency virus (HIV) who have CD4+ T-cell counts >= 350 cells/uL and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections in the last year are allowed
* Willingness to undergo mandatory pre-treatment biopsy (unless there is adequate archival tumor specimen available for PD-L1 IHC evaluation)
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Or, female subjects of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first study drug administration
* Male and female subjects who are of reproductive potential must agree to use highly effective method of birth control (e.g., implants, injectables, birth control pills with two hormones, intrauterine devices [IUDs], complete abstinence or sterilized partner, and female sterilization) and a barrier method (e.g., condoms, vaginal ring, sponge, etc.) during the period of therapy and for 4 months after the last dose of study drug
* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements
* Must be able to swallow study drug

Exclusion Criteria:

* Receiving radiation =< 14 days prior to enrollment to the site of selected target lesions
* Systemic therapy for cancer =< 21 days prior to enrollment
* Autoimmune disorder requiring active therapy as defined by corticosteroids at a dose >= 10 mg oral prednisone or the equivalent or requiring chronic immunosuppressive therapy
* Use of corticosteroids =< 14 days prior to enrollment at a dose of >= 10 mg oral prednisone or the equivalent per day
* Received immune checkpoint inhibitor therapy (anti-PD-1, anti-PD-L1, or anti-CTLA4 directed therapy) on a prior clinical trial
* Has received selinexor or another XPO1 inhibitor previously
* Any active gastrointestinal dysfunction that could interfere with absorption of study treatment in the opinion of the investigator
* Pregnant or lactating women
* Any condition that would prohibit the understanding or rendering of informed consent
* Any condition including additional malignancies, laboratory abnormalities, or psychiatric illness that in the opinion of the investigator would interfere with the patient's safety or compliance while on trial
* Severe infection that in the opinion of the investigator would interfere with patient safety or compliance on trial within 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated prior to patients being enrolled at the second dose level.
Groups:
- Treatment (Selinexor, Pembrolizumab): Patients received study intervention at Dose Level 1 (starting dose): selinexor 80mg PO on days 1, 8 and 15, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity. Pembrolizumab: Given IV. Selinexor: Given PO.
  No patients enrolled at other dose levels,
Period: Overall Study
Arm/Group | Treatment (Selinexor, Pembrolizumab)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Selinexor, Pembrolizumab): Patients receive selinexor PO on days 1, 8 and 15, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity. Pembrolizumab: Given IV. Selinexor: Given PO
Arm/Group | Treatment (Selinexor, Pembrolizumab)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) (Phase Ib)
Description: Defined by dose-limiting toxicity (DLTs). Dose limiting toxicities will be listed according to dose level. Separately by dose level and the expansion cohort (as well as for the total RP2D cohort), adverse events (AEs) will be summarized as number of patients according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 term and grade, where grade is the maximum across a patient's treatment period.
Time Frame: Up to 2 cycles (each cycle is 21 days); up to about 6 weeks
Population: 3 patients treated at dose level 1 were evaluable before study was terminated.
Measure: Number; unit: mg Selinexor
Groups:
- Treatment (Selinexor, Pembrolizumab): Patients receive selinexor PO on days 1, 8 and 15, and pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 21 days for 24 months in the absence of disease progression or unacceptable toxicity.
  Pembrolizumab: 200 mg, given IV
  Selinexor: 80 mg, given PO
Arm/Group | Treatment (Selinexor, Pembrolizumab)
Number analyzed (Participants) | 3
mg Selinexor | NA — Study was terminated prematurely, and insufficient number of patients were enrolled to assess this outcome measure.

2. Primary Outcome: Objective Response Rate (ORR) (Phase II)
Description: ORR, calculated as the total number of patients with a confirmed complete response or partial response, will be reported as a percentage of total evaluable patients. Response will be reported using Response Evaluation Criteria in Solid Tumor 1.1 definitions. ORR will be summarized by exact binomial 95% confidence intervals (CI).
Time Frame: Up to approximately 2 years 4 months
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Selinexor, Pembrolizumab)
Number analyzed (Participants) | 4
percentage of patients | 75

3. Secondary Outcome: Number of Patients Who Experience a Grade 3 or Higher Adverse Event (AE).
Description: Defined by NCI CTCAE version 5. The number of patients who experience at least one grade 3-5 AEs will be reported.
Time Frame: Up to approximately 1 year 7 months.
Population: 4 patients were enrolled, after which study was terminated; 4 patients were evaluable for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Selinexor, Pembrolizumab)
Number analyzed (Participants) | 4
Participants | 1

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as the median time from initiation of study intervention to progressive disease, defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0).
Time Frame: From enrollment to trial to time of disease progression or death from any cause, assessed up to 2 year 4 months.
Measure: Mean (Full Range); unit: months
Arm/Group | Treatment (Selinexor, Pembrolizumab)
Number analyzed (Participants) | 4
months | NA [0 to NA] — Median PFS not determined because PFS was not reached by any patient (0 to not reached) at the time of data cut-off due to the study being prematurely terminated.

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events assessed from first dose to 30 days after last treatment, approximately up to 1 year 7 months. All-cause mortality assessed from enrollment until death from any cause, approximately 2 years 4 months.
Arm/Group | Treatment (Selinexor, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selinexor, Pembrolizumab) (N=4)
Sepsis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Selinexor, Pembrolizumab) (N=4)
Abdominal pain (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood bicarbonate decreased (Investigations) | 2
Blurred vision (Eye disorders) | 2
Cataract (Eye disorders) | 2
Chills (General disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 2
Dry eye (Eye disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fullness in ears (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Gritty eyes (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 2
Floaters (Eye disorders) | 1
Generalized edema (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
COVID 19 (Infections and infestations) | 1
Flu (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 1
Lymphocyte count decreased (Investigations) | 3
Malaise (General disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Neck edema (General disorders) | 1
Neutrophil count decreased (Investigations) | 3
Non-cardiac chest pain (Gastrointestinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Platelet count decreased (Investigations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other: Hallux great toe (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other: Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other: Lip lesion (discoloration) (Skin and subcutaneous tissue disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04856189/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT04856189/ICF_001.pdf